CLINICAL TRIAL: NCT04842760
Title: PLATELET Function Assay With Flow Imaging on ImageSTREAM Cytometer
Acronym: PLATELETSTREAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0039
Record Dates: First submitted 2021-04-07; First posted 2021-04-13 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Platelet Disorder; Heparin-induced Thrombocytopenia; Platelet Activation; Platelet Aggregation
Keywords: Platelet Disorder; Heparin-induced Thrombocytopenia; ImageStream cytometer; Platelet activation; Platelet aggregation
MeSH Terms: conditions — Blood Platelet Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No platelet disorders or no HIT: Patients without platelet disorders or without HIT, without anti-PF4/H antibodies, without anti-aggregant treatment.
- HIT patients with anti-PF4/H antibodies: patients with anti-PF4/H antibodies but for whom HIT was ruled out.
- platelet dysfunction or HIT: Patients with platelet dysfunction or suffering from HIT

SUMMARY:
Platelets are essential blood elements to maintain hemostasis. Quantitative or qualitative defects can be responsible of hemorrhagic (platelet disorders) or thrombotic (heparin induced thrombocytopenia [HIT]) troubles. Diagnosis of these pathologies is sometimes urgent and consists in delicate platelet functional assays that are mostly made in expert centers. These platelets functional assays measure platelets activation and/or aggregation in response to diverse inductors and may lack sensitivity. The investigators would like to propose a new diagnostic tool with the use of imaging flow cytometry which provides much more information than classic cytometer on cell morphology thanks to images collected by the optical channel of the ImageStream cytometer. The use of this cytometer offers an innovative approach.

This study is a monocentric prospective and non-interventional study. The investigators will analyze patient samples with the ImageStream cytometer and reference laboratory tests (light transmission aggregometry and serotonin release assay) in parallel and compare results from the different techniques. This new diagnostic technique will demonstrate a non-inferiority diagnosis compared to reference tests and maybe a better sensibility.

ELIGIBILITY:
Inclusion Criteria:

* male or female patient for whom a blood test was prescribed in a context of diagnosis of platelet dysfunction or HIT

Exclusion Criteria:

* minor patients
* patients who have opposed the use of their personal data for research work.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male or female patient for whom a blood test was prescribed in a context of diagnosis of platelet dysfunction or HIT.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Concordance between ImageStream cytometer and reference laboratory tests for platelet disorders diagnosis | 12 months
  platelet disorders reference laboratory tests are light transmission aggregometry and serotonin release assay
Concordance between ImageStream cytometer and reference laboratory tests for HIT diagnosis | 12 months
  reference laboratory tests are light transmission aggregometry and serotonin release assay

SECONDARY OUTCOMES:
Characterization of platelet morphology with ImageStream | 12 months
  Analyses of data provided by the ImageStream system on platelets and platelets aggregates

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No